CLINICAL TRIAL: NCT03136757
Title: Analysis of Transcriptomic Profile of Graft-versus-host Disease (GHVD) After Allogeneic Grafting of Hematopoietic Stem Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2016_843_0016
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Graft Vs Host Disease; Hematopoietic Stem Cells
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Transcriptomic analysis of GVHD biopsies — The transcriptomic analysis of GVHD biopsies aims at:
  * to demonstrate an evocative or even specific molecular profile, making the diagnosis of GVHD easier
  * to identify new intracellular signaling pathways that could lead to new therapeutic

SUMMARY:
Graft-versus-host disease (GVHD) is a frequent and severe complication of hematopoietic stem cell transplantation (HSC), and is responsible for significant early mortality despite prophylactic strategies developed in recent decades, Especially since it is resistant to first-line treatment.

The present diagnosis is difficult, non-specific and is based on the combination of an evocative clinical context (CSH allograft, time to appearance before J100, characteristic clinical manifestations), suggestive anatomo-pathological analysis (predominantly inflammatory infiltrate Lymphocyte, mucosal edema and presence of apoptotic bodies), and the exclusion of any differential diagnosis (in particular serology / negative viral PCR).

However, to date there is no molecular characterization of this manifestation, and therefore no specific treatment.

The nCounter® nanostring technology allows the rapid and simple analysis of the simultaneous expression of a group of genes (up to 800 on the same sample), from a very small amount of RNA, and from samples with difficulty Such as fabrics already fixed to formaldehyde and included in paraffin. It allows the detection of a "molecular signature" of the tissue analyzed.

No transcriptomic analysis has ever been performed on human tissues with GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Person aged ≥ 18 years
* Patients who have received an HSC allograft since June 2012
* Having presented a suspicion of cutaneous or digestive GVHD before J100 post-allograft
* Of which the diagnosis was retained by the combination of clinical and histological criteria
* Or whose diagnosis has been reversed by histological analysis, for the reactive / inflammatory biopsies that serve as control
* The diagnosis of which was made between 01/01/2013 and 31/12/2015
* Survived at least 1 month to monitor clinical progress

Exclusion Criteria:

* Whose biopsy specimens were also the sites of a viral reactivation (EBV, CMV, HHV) that could mimic a GVHD
* Having survived less than 1 month after the diagnosis of GVHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recovery of fixed and paraffin-embedded biopsy fragments previously performed during the diagnosis of GVHD, not used for routine histological analysis because in excess, and stored in the pathology laboratory
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-08-20 (Estimated); Primary Completion 2017-10-20 (Estimated); Study Completion 2017-10-20 (Estimated)

PRIMARY OUTCOMES:
Transcriptomic profile by analysis of the expression of the mRNAs of a determined panel of 800 genes regulating the immune response | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France